CLINICAL TRIAL: NCT01975350
Title: Prospective Observation of Colistimethate Sodium Inhalation in Patients With Ventilator-associated Tracheobronchitis/Pneumonia or Lower Respiratory Tract Colonization by Multidrug Resistant Gram-negative Bacteria
Brief Title: Efficacy Study of Colistimethate Sodium Inhalation in Patients With Ventilator-associated Pneumonia
Status: Terminated | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201303119MINB
Record Dates: First submitted 2013-10-22; First posted 2013-11-04 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2013-10

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Colistimethate sodium inhalation
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Colistimethate sodium inhalation: Colistimethate sodium inhalation for patients with ventilator-associated tracheobronchitis, pneumonia or lower respiratory tract colonization by multidrug resistant Gram-negative bacteria.
  Additional intravenous colistimethate sodium for patients with ventilator-associated pneumonia
- saline inhalation: saline inhalation for patients with ventilator-associated tracheobronchitis, pneumonia or lower respiratory tract colonization by multidrug resistant Gram-negative bacteria.

SUMMARY:
There might be additional benefit on clinical outcomes from adjunctive colistimethate sodium inhalation as therapy for multidrug resistant Gram-negative ventilator-associated pneumonia.

DETAILED DESCRIPTION:
Besides, early antibiotics intervention might be benefit for patients with ventilator-associated tracheobronchitis or lower airway colonization with multidrug resistant Gram-negative bacteria.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 20 years old
2. medical ICU patients with invasive ventilator use ≥ 48 hours
3. multidrug resistant Gram-negative bacteria obtained from lower respiratory tract

Exclusion Criteria:

1. pregnancy
2. concurrent use of other antimicrobial agents active for isolated multidrug resistant Gram-negative bacteria (as defined as resistant to carbapenem, fluoroquinolone, and anti-pseudomonas beta-lactams), such as tigecycline, aminoglycosides, and sulbactam
3. patients who refuse to receive any inhaled therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in medical intensive care unit with ventilator use
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2013-10-01; Primary Completion 2016-02-04 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
clinical cure rate | From date of starting colistimethate sodium to 28th days or til discharge from hospital, whichever came first, assessed up to 28 days
  including clinical improvement and microbiological outcome(eradication of the pathogen as no growth of the pathogen in the final culture of specimens during the entire hospitalization)

SECONDARY OUTCOMES:
intensive care unit stay | From date of starting colistimethate sodium to discharge date of intensive care unit, assessed up to 3 months
hospital stay | From date of starting colistimethate sodium to discharge date of hospital, assessed up to 3 months
all cause mortality | From date of starting colistimethate sodium to 28th days or til death, whichever came first, assessed up to 28 days
ventilator-associated pneumonia-related mortality | Death that occurred during the colistimethate sodium treatment period when the signs of pneumonia remained and as death due to septic shock, assessed up to 28 days
microbiologic eradication in colonization patients | From date of starting colistimethate sodium to 28th days or til discharge from hospital, whichever came first, assessed up to 28 days
ventilator-associated pneumonia rate | From date of starting colistimethate sodium to discharge date of hospital, assessed up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wang-Huei Sheng, M.D. Ph.D, Principal Investigator — Center of Infection Control of National University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan